CLINICAL TRIAL: NCT01672073
Title: An Open, Non-randomised, Study to Provide Data on the Arterial Pressure Wave Form Obtained Through the Proxima 3 in Patients Who Require the Insertion of an Arterial Line
Brief Title: Analysis of the Arterial Pressure Wave Form Through the Proxima Device
Status: Completed | Type: Observational
Sponsor: Sphere Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROX005
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Local Pressure Effects
Keywords: pressure; waveform; arterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the trial is to confirm that the presence of the Proxima 3 disposable in the arterial line doesn't significantly attenuate the arterial pressure wave form. The principal aim of the trial will be:

• To obtain quantitative data allowing investigation of the pressure wave form obtained in a standard arterial line compared to various arterial lines fitted with the Proxima 3.

DETAILED DESCRIPTION:
The purpose of this study is to examine the transmission of the arterial pressure wave form through Proxima 3 disposable attached to a configurable parts of the patient's arterial line. The Proxima device has been tested by Intertek as part of the Proxima 2 project and found to comply to BS EN 60601-1 2nd edition "Medical electrical equipment - Part 1: General requirements for basic safety and essential performance". Additional internal tests have also been carried out for clause 51.103, frequency response, from BS EN 60601-2-34(2001).

This study part of the on-going development of the Proxima system which monitors metabolic parameters in critically ill patients using a disposable sensor array. This study builds upon the four clinical trials carried out in the past two years by Sphere Medical in partnership with the NHS (REC references: 10/H1308/53, 10/H0308/113, 11/SW/0166, 12/SW/0175).

This study forms part of the development process for the Proxima family of devices.

The Proxima 3:

* Is a disposable multi-parameter microanalyser
* Is connected into the patient's arterial line.
* Will measure all or some of blood gases, haematocrit and electrolytes and is connected to a small bedside monitor, which displays the results.
* Microanalyser can perform an unlimited number of analyses over a period of up to seventy two hours.
* Will be used as part of a closed system, reducing infection risk and preventing blood loss.

Proxima 3 will enable clinicians to measure blood parameters without leaving the patient's bedside. This will support the ability to respond rapidly to changing conditions in their critically ill patients. The measurements made by the Proxima 3 system have the potential to inform clinical decision support systems and to change, at a fundamental level, the ability of clinicians to improve patient care.

In this study the Proxima 3 is a passive component. It will NOT be connected to the Proxima 3 monitor. NO blood will be taken and NO analysis of the blood analyte concentrations will occur in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 18
* Patients will give full informed consent to participate in the study before inclusion.
* All patients who have an arterial line inserted as standard care will be considered for inclusion.

Exclusion Criteria:

* Refusal of consent to participate
* The patient is considered by the investigator to be unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Intensive Care or High Dependency Units who require an arterial line to be inserted as standard care
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To confirm that siting Proxima 3 in the arterial line does not affect the pressure wave form | 10 minutes maximum
  The data traces collected from the arterial pressure waveform monitor will undergo quantitative assessment to determine the effect on the pressure wave, if any, by introducing the Proxima 3 device in the system.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clutton-Brock, MB ChB FRCP, Study Director — Queen Elizabeth Hopsital, Birmingham, UK
Locations (1):
- Queen Elizabeth Hospital, City and Borough of Birmingham, Edgbaston, United Kingdom

REFERENCES:
- See also: Click here for more information about this study — http://www.spheremedical.com